CLINICAL TRIAL: NCT03530124
Title: A Prospective, Randomized, Open-label Clinical Trial to Assess Apnea Following Administration of 13-valent Conjugate Pneumococcal Vaccine, Diphtheria Toxoid, Tetanus Toxoid, and Acellular Pertussis Vaccine, Inactivated Polio Vaccine, Hepatitis B Vaccine, and Haemophilus Influenzae Type B Vaccine in Preterm Infants
Brief Title: Apnea in Hospitalized Preterm Infants Following the Administration of Routine Childhood Vaccines
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: Centers for Disease Control and Prevention (U.S. Federal Agency); Children's Hospital Medical Center, Cincinnati (Other); University of North Carolina (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: Pro00088094; 200 2012 53663 0010 (Other Grant/Funding Number: CDC)
Record Dates: First submitted 2018-05-08; First posted 2018-05-21 (Actual); Results first posted 2023-01-11 (Actual); Last update posted 2024-02-14 (Actual); Status verified 2024-02

CONDITIONS: Apnea; Apnea Neonatal; Prematurity
Keywords: apnea following vaccination
MeSH Terms: conditions — Apnea; Premature Birth | interventions — Diphtheria-Tetanus-acellular Pertussis Vaccines; Hepatitis B Vaccines; Poliovirus Vaccine, Inactivated

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Vaccinated (Other): In the study arm, infants will receive PCV13, DTaP, HBV, IPV, and Hib vaccines within 12 hours of randomization. Infants will be monitored from time of vaccination to 48 hours post-vaccination for the occurrence of apnea, bradycardia and desaturation.
  Interventions: Biological: PCV13; Biological: DTaP; Biological: HBV; Biological: IPV; Biological: Hib
- Unvaccinated (No Intervention): In the study arm, infants will not receive PCV13, DTaP, HBV, IPV, and Hib vaccines during the study. Infants will be monitored from randomization to 48 hours post-randomization for the occurrence of apnea, bradycardia and desaturation.

INTERVENTIONS:
Biological: PCV13 — Advisory Committee on Immunization Practices (ACIP) Recommended vaccine
  Other Names: 13-valent Conjugate Pneumococcal Vaccine
  Arms: Vaccinated
Biological: DTaP — ACIP Recommended vaccine
  Other Names: Diphtheria, Tetanus, and Acellular Pertussis Vaccine
  Arms: Vaccinated
Biological: HBV — ACIP Recommended vaccine
  Other Names: Hepatitis B Vaccine
  Arms: Vaccinated
Biological: IPV — ACIP Recommended vaccine
  Other Names: Inactivated Polio Vaccine
  Arms: Vaccinated
Biological: Hib — ACIP Recommended vaccine
  Other Names: Haemophilus influenzae Type B Vaccine
  Arms: Vaccinated

SUMMARY:
A prospective, randomized open-label clinical trial will be conducted from July 2018 to October 2020. Approximately 300 preterm infants will be enrolled across three sites: Duke University Medical Center, the University of North Carolina, and Cincinnati Children's Hospital Medical Center. Eligible infants will be randomized 1:1 to receive either 2-month US licensed childhood vaccines (PCV13, DTaP, HBV, IPV an Hib) or no vaccines. After their participation in the study, healthcare providers of the infants in the unvaccinated group will make decision abut receipt of their 2-month childhood vaccines. The study will collect data from the continuous cardiorespiratory and pulse oximetry monitors from randomization to 48 hours after randomization for infants in the unvaccinated group, and from randomization to 48 hours after vaccination for infants in the vaccinated group. Infants in both groups will be monitored for up to 60 hours for the occurrence of apnea, bradycardia, and oxygen desaturation. For infants in the "vaccinated" group, the study will also collect adverse events of clinical interest and serious adverse events occurring between the end of the 48-hour monitoring period and 14 days after vaccination. This information will be collected through parental report and review of medical records.

DETAILED DESCRIPTION:
Modified Intent-to-Treat (mITT) Analysis Population: Defined as any infant that was enrolled and randomized in the study

For the mITT analysis, infants will be analyzed in their assigned treatment arms irrespective of receipt of vaccine. Study outcomes will be included in the analysis as follows:

i) Vaccinated group: study outcomes in the 48-hour monitoring after vaccination. If vaccination does not occur by 12 hours after randomization, then study outcomes will be assessed between 12 and 60 hours after randomization.

ii) Unvaccinated group: study outcomes in the 48-hour monitoring period after randomization.

ELIGIBILITY:
Inclusion Criteria:

1. <33 and 0 days weeks gestational age at birth
2. ≥6 weeks and 0 days and ≤12 weeks and 0 days postnatal age at randomization
3. Remains hospitalized after birth (has never been discharged home)
4. Treating clinician deems infant eligible to receive 2-month vaccines
5. English- or Spanish-speaking parent(s)/legally authorized representative(s) (LAR(s))
6. Not planned for discharge within 60 hours of study entry
7. The parent/guardian must be willing and capable of providing permission for their child to participate through the written informed consent process

Exclusion Criteria:

1. Receipt of DTaP, IPV, PCV13, or Hib prior to enrollment. Previous administration of the first dose of HBV is permitted
2. Anticipated receipt of any vaccine other than DTaP, IPV, HBV, PCV13, or Hib during the first 60 hours after randomization
3. History of a severe allergic reaction (e.g. anaphylaxis) to a previous dose of any hepatitis B vaccine
4. History of a severe allergic reaction (e.g. anaphylaxis) to any component of the vaccines used in the study including neomycin, yeast and polymyxin B
5. History of latex allergy
6. Fever ≥38°C within 48 hours prior to randomization*

   *This may result in a temporary delay of randomization
7. Active known respiratory infection within 48 hours prior to randomization*

   *This may result in a temporary delay of randomization
8. Active infection being treated with systemic antimicrobials*

   *This may result in a temporary delay of randomization
9. Requiring mechanical ventilation or support with nasal intermittent positive pressure ventilation (NIPPV)*

   *This may result in a temporary delay of randomization
10. History of unstable progressive neurologic disorder of unknown cause
11. Known cause of apnea other than apnea of prematurity
12. Cyanotic heart disease (congenital or acquired)
13. Major invasive medical or surgical procedure (including circumcision) within 48 hours prior to randomization or anticipated to have major invasive medical or surgical procedure during the first 60 hours after randomization*

    *This may result in a temporary delay of randomization
14. Child or parent/LAR is an immediate relative of study staff or an employee who is supervised by study staff.
15. Any condition that would, in the opinion of the site investigator, place the participant at an unacceptable risk of injury or render the participant unable to meet the requirements of the protocol

Min Age: 6 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 223 (Actual)
Dates: Start 2018-07-17 (Actual); Primary Completion 2021-11-01 (Actual); Study Completion 2021-11-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rachel G Greenberg, MD, Principal Investigator — Duke University; Andrea Trembath, MD, Principal Investigator — University of North Carolina; Mary A Staat, MD, Principal Investigator — Children's Hospital Medical Center, Cincinnati; Karen Broder, MD, Principal Investigator — Centers for Disease Control and Prevention
Locations (4):
- United States (4):
  - Centers for Disease Control and Prevention, Atlanta, Georgia
  - University of North Carolina, Chapel Hill, North Carolina
  - Duke University, Durham, North Carolina
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Greenberg RG, Rountree W, Staat MA, Schlaudecker EP, Poindexter B, Trembath A, Laughon M, Poniewierski MS, Spreng RL, Broder KR, Wodi AP, Museru O, Anyalechi EG, Marquez PL, Randolph EA, Aleem S, Kilpatrick R, Walter EB. Apnea After 2-Month Vaccinations in Hospitalized Preterm Infants: A Randomized Clinical Trial. JAMA Pediatr. 2025 Mar 1;179(3):246-254. doi: 10.1001/jamapediatrics.2024.5311. PMID 39761016

RESULTS

PARTICIPANT FLOW:
Groups:
- Vaccinated: In the study arm, infants will receive PCV13, DTaP, HBV, IPV, and Hib vaccines within 12 hours of randomization. Infants will be monitored from time of vaccination to 48 hours post-vaccination for the occurrence of apnea, bradycardia and desaturation.
  PCV13: ACIP Recommended vaccine
  DTaP: ACIP Recommended vaccine
  HBV: ACIP Recommended vaccine
  IPV: ACIP Recommended vaccine
  Hib: ACIP Recommended vaccine
Period: Overall Study
Arm/Group | Vaccinated | Unvaccinated
Started | 107 | 116
Completed | 105 | 115
Not Completed | 2 | 1
Not completed — Withdrawal by Subject | 0 | 1
Not completed — Protocol Violation | 1 | 0
Not completed — Discharged prior to study completion | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Vaccinated | Unvaccinated | Total
Number analyzed (Participants) | 107 | 116 | 223
Age, Continuous [Median (Full Range); unit: Gestational Age in Weeks]
  Gestational Age at Birth | 27.3 [23.0 to 32.9] | 27.7 [23.0 to 32.7] | 27.6 [23.0 to 32.9]
Age, Customized [Count of Participants; unit: Participants] — Gestational Age in Weeks
  Participants
    Age: <28 wks | 60 | 61 | 121
    Age: >=28 wks | 47 | 55 | 102
Age, Customized [Median (Full Range); unit: Postmenstrual Age in Weeks] — Postmenstrual age is defined as the sum of gestational age plus postnatal age
  Postmenstrual Age in Weeks
    Postmenstrual Age | 36.6 [32.0 to 42.0] | 36.6 [32.4 to 43.6] | 36.6 [32.0 to 43.6]
Age, Customized [Median (Full Range); unit: Postnatal Age in Weeks]
  Postnatal Age | 8.7 [6.4 to 11.9] | 8.7 [6.3 to 12.0] | 8.7 [6.3 to 12.0]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 57 | 60 | 117
  Male | 50 | 56 | 106
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 16 | 10 | 26
  Not Hispanic or Latino | 89 | 103 | 192
  Unknown or Not Reported | 2 | 3 | 5
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White Only | 55 | 66 | 121
  Black Only | 33 | 42 | 75
  Other | 19 | 8 | 27
Multiple Gestation [Count of Participants; unit: Participants]
  Single | 73 | 84 | 157
  Twins | 34 | 30 | 64
  Triplets | 0 | 2 | 2
Birth Weight [Median (Full Range); unit: Grams] | 940 [449 to 2860] | 1000 [430 to 2550] | 970 [430 to 2860]
Insurance [Count of Participants; unit: Participants]
  Any Private | 50 | 49 | 99
  Public | 55 | 66 | 121
  None | 2 | 1 | 3
Reason for Preterm Delivery [Count of Participants; unit: Participants]
  Hypertension/Preeclampsia/Hemolysis, Elevated Liver Enzymes, Low Platelet Count (HELLP) | 30 | 25 | 55
  Preterm Labor/Premature Rupture | 55 | 69 | 124
  Placental Abruption | 12 | 12 | 24
  Fetal distress | 18 | 22 | 40
  Other | 25 | 29 | 54
Received Synagis During Study Period [Count of Participants; unit: Participants]
  Yes | 0 | 1 | 1
  No | 107 | 115 | 222
Received Caffeine [Count of Participants; unit: Participants] — Population: Data not collected on 6 participants.
  Participants
    number analyzed (Participants) | 102 | 115 | 217
    Yes | 98 | 107 | 205
    No | 4 | 8 | 12
Sibling Enrolled in Study [Count of Participants; unit: Participants]
  Yes | 28 | 24 | 52
  No | 79 | 92 | 171
Respiratory Support at Randomization [Count of Participants; unit: Participants] — Population: Data not collected on 1 participant.
  Participants
    number analyzed (Participants) | 106 | 116 | 222
    Continuous Positive Airway Pressure (CPAP) | 17 | 16 | 33
    Nasal Cannula | 34 | 46 | 80
    None | 55 | 54 | 109
Combination Vaccine Brand Administered [Count of Participants; unit: Participants] — Pediarix contains DTap-IPV-HBV; Pentacel contains DTaP-IPV-Hib Population: Collection of combination vaccine data were collected for the vaccinated arm only. Data not collected on 5 participants.
  Participants
    Pediarix: number analyzed (Participants) | 102 | 0 | 102
    Pediarix | 100 | 0 | 100
    Pentacel: number analyzed (Participants) | 102 | 0 | 102
    Pentacel | 2 | 0 | 2
Haemophilus influenzae type b Vaccine Brand Administered [Count of Participants; unit: Participants] — Population: Collection of Haemophilus influenzae type b vaccine data were collected for the vaccinated arm only. Data not collected on 7 participants.
  Participants
    ActHIB: number analyzed (Participants) | 100 | 0 | 100
    ActHIB | 98 | 0 | 98
    PedvaxHIB: number analyzed (Participants) | 100 | 0 | 100
    PedvaxHIB | 1 | 0 | 1
    Hiberix: number analyzed (Participants) | 100 | 0 | 100
    Hiberix | 1 | 0 | 1
Hepatitis B Vaccine Brand Administered - Engerix-B [Count of Participants; unit: Participants] — Engerix-B is the only Hepatitis B vaccine reported during study period Population: Collection of Hepatitis B vaccine data were collected for the vaccinated arm only.
  Participants
    number analyzed (Participants) | 107 | 0 | 107
    (all) | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Occurrence of Apnea
Description: Number of infants with ≥ 1 apneic event in a 48-hour monitoring period after vaccination in the "vaccinated" group and a 48-hour monitoring period after randomization in the "unvaccinated" group, mITT Population
  Apnea was defined as a pause in respirations of >20 seconds, or a pause in respirations of >15 seconds with associated bradycardia (heart rate <80 beats per minute for any duration occurring within 1 minute of the apnea event). Potential apnea events triggered by the cardiorespiratory monitors were manually reviewed by 2 neonatologists to verify the event. In uncommon situations in which manual review of a triggered event was not possible due to missing data, the triggered event was considered to be apnea.
Time Frame: 48 hours
Population: The mITT population includes any infant that was enrolled and randomized in the study.
Measure: Count of Participants; unit: Participants
Arm/Group | Vaccinated | Unvaccinated
Number analyzed (Participants) | 107 | 116
Participants
  Yes | 25 | 12
  No | 80 | 104
  Missing | 2 | 0
Statistical Analysis 1: Comparison: Vaccinated vs Unvaccinated; Test type: Superiority — The number of infants with ≥1 apneic event for each group and compared using a Mantel-Haenszel statistic in a stratified analysis by study site and gestational age group (< 28 weeks versus ≥ 28 weeks) to control for the randomization blocks at the two-sided alpha 0.05 level and corresponding 95% confidence interval for the occurrence of apnea; p = 0.0104, Mantel Haenszel; Odds Ratio (OR) = 2.70, 95% CI 2-sided [1.27 to 5.73] — No adjustments were made to the alpha level (two-sided alpha=0.05) for the primary objective

2. Secondary Outcome: Number of Apneic Episodes
Description: Average number of apneic episodes in a 48-hour monitoring period after vaccination in the "vaccinated" group and a 48-hour monitoring period after randomization in the "unvaccinated" group.
Time Frame: 48 hours
Population: The mITT population includes any infant that was enrolled and randomized in the study.
Measure: Mean (Standard Deviation); unit: Apneic Episodes
Arm/Group | Vaccinated | Unvaccinated
Number analyzed (Participants) | 107 | 116
Apneic Episodes | 2.72 (2.76) | 2.00 (1.76)
Statistical Analysis 1: Comparison: Vaccinated vs Unvaccinated; Test type: Other — The number of apnea events were compared using a linear regression model (assuming a Poisson distribution) with study site and gestational age group covariates to control for the randomization blocks; p = 0.11, Regression, Linear; No adjustments were made to the alpha level (two-sided alpha=0.05) for the secondary objectives

3. Secondary Outcome: Duration of Apneic Episodes
Description: Average duration of apneic episodes in a 48-hour monitoring period after vaccination in the "vaccinated" group and a 48-hour monitoring period after randomization in the "unvaccinated" group.
Time Frame: 48 hours
Population: The mITT population includes any infant that was enrolled and randomized in the study.
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Vaccinated | Unvaccinated
Number analyzed (Participants) | 107 | 116
seconds | 27.7 (2.6) | 32.3 (4.7)
Statistical Analysis 1: Comparison: Vaccinated vs Unvaccinated; Test type: Other — Average duration of apnea episodes between groups were compared using a mixed effects model with a random intercept for each infant with one or more events and study site and gestational age group as covariates to control for the randomization blocks; p = 0.36, Mixed Effects Model; No adjustments were made to the alpha level (two-sided alpha=0.05) for the secondary objectives

4. Secondary Outcome: Increase in Respiratory Support
Description: Proportion of infants requiring any increase in respiratory support in a 48-hour monitoring period after vaccination in the "vaccinated" group and a 48-hour monitoring period after randomization in the "unvaccinated" group.
Time Frame: 48 hours
Population: The mITT population includes any infant that was enrolled and randomized in the study.
Measure: Count of Participants; unit: Participants
Arm/Group | Vaccinated | Unvaccinated
Number analyzed (Participants) | 107 | 116
Participants
  Yes | 8 | 4
  No | 92 | 112
  Missing | 7 | 0
Statistical Analysis 1: Comparison: Vaccinated vs Unvaccinated; Test type: Superiority — The proportion of infants requiring an increase in respiratory support for each group were compared using a Mantel-Haenszel statistic in a stratified analysis by study site and gestational age group to control for the randomization blocks at the two-sided alpha 0.05 level and corresponding 95% confidence interval for the occurrence of apnea; p = 0.3555, Mantel Haenszel; Odds Ratio (OR) = 2.07, 95% CI 2-sided [0.59 to 7.23] — No adjustments were made to the alpha level (two-sided alpha=0.05) for the secondary objectives

5. Secondary Outcome: Severe Cardiorespiratory Events
Description: Proportion of infants with severe ≥1 severe cardiorespiratory event in a 48-hour monitoring period after vaccination in the "vaccinated" group and a 48-hour monitoring period after randomization in the "unvaccinated" group.
  Only severe apnea events in the mITT analysis window and only the severe bradycardia events in the mITT analysis window from Duke University. The monitor data were not viable at UNC and Cincinnati Children's Hospital. Duke data were adjudicated by neonatologists.
Time Frame: 48 hours
Population: mITT Analysis Population: Duke Site Only
Measure: Count of Participants; unit: Participants
Arm/Group | Vaccinated | Unvaccinated
Number analyzed (Participants) | 39 | 42
Participants
  Yes | 7 | 8
  No | 31 | 34
  Missing | 1 | 0
Statistical Analysis 1: Comparison: Vaccinated vs Unvaccinated; Only Duke University had viable monitoring data to analyze this compound outcome objective; Test type: Superiority — The proportion of infants with ≥1 cardiorespiratory event using a Mantel-Haenszel statistic in at the two-sided alpha 0.05 level and corresponding 95% confidence interval; p = 1.0000, Mantel Haenszel; Odds Ratio (OR) = 0.89, 95% CI 2-sided [0.29 to 2.77] — No adjustments were made to the alpha level (two-sided alpha=0.05) for the secondary objectives

6. Secondary Outcome: Positive Pressure Ventilation
Description: Proportion of Infants Requiring Positive Pressure Ventilation in a 48-hour monitoring period after vaccination in the "vaccinated" group and a 48-hour monitoring period after randomization in the "unvaccinated" group.
Time Frame: 48 hours
Population: The mITT population includes any infant that was enrolled and randomized in the study.
Measure: Count of Participants; unit: Participants
Arm/Group | Vaccinated | Unvaccinated
Number analyzed (Participants) | 107 | 116
Participants
  Yes | 2 | 1
  No | 104 | 115
  Missing | 1 | 0
Statistical Analysis 1: Comparison: Vaccinated vs Unvaccinated; The proportion of infants requiring positive pressure ventilation for each group were compared using a Mantel-Haenszel statistic in a stratified analysis by study site and gestational age group to control for the randomization blocks at the two-sided alpha 0.05 level and corresponding 95% confidence interval for the occurrence of apnea during the 48-hour monitoring period; Test type: Superiority; p = 1.0000, Mantel Haenszel; Odds Ratio (OR) = 1.93, 95% CI 2-sided [0.17 to 21.63] — No adjustments were made to the alpha level (two-sided alpha=0.05) for the secondary objectives

ADVERSE EVENTS:
Time Frame: Unvaccinated infants and vaccinated infants were followed for 48 hours for clinically important adverse events and serious adverse events. In addition, vaccinated infants were followed for 14 days after vaccination for clinically important adverse events and serious adverse events.
Description: All clinically important adverse events (not including serious adverse event) outcome data were reported out within the study outcome measures.
Arm/Group | Vaccinated | Unvaccinated
All-Cause Mortality (participants affected / at risk) | 0/107 | 0/116
Serious Adverse Events (participants affected / at risk) | 1/107 | 0/116
Other Adverse Events (participants affected / at risk) | 32/107 | 20/116
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Vaccinated (N=107) | Unvaccinated (N=116)
Hospital readmission for tachypnea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Hospital readmission for retinopathy of prematurity (Eye disorders) | 1 (1) | 0 (0)
Respiratory decompensation and hypotension following elective surgery (Surgical and medical procedures) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Vaccinated (N=107) | Unvaccinated (N=116)
Severe Cardiorespiratory Event (Cardiac disorders) | 7/39 (39) | 8/42 (8) — Severe cardiorespiratory events were defined according to the protocol. Definition: Respiratory pause of >30 seconds in duration or bradycardia of <60 beats per minute for >10 seconds Duke Site Only - See Secondary Outcome #5
≥ 1 Apneic Event (Respiratory, thoracic and mediastinal disorders) | 25 (25) | 12 (12) — Apneic events were defined according to the protocol. Definition: A pause in respirations of >20 seconds, or a pause in respirations of >15 seconds with associated bradycardia (heart rate <80 beats per minute) -See Primary Outcome #1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2024-01-22): https://cdn.clinicaltrials.gov/large-docs/24/NCT03530124/Prot_002.pdf
  • Statistical Analysis Plan (2022-10-14): https://cdn.clinicaltrials.gov/large-docs/24/NCT03530124/SAP_001.pdf